CLINICAL TRIAL: NCT06939218
Title: Analysis of New Materials and Artificial Turf Products: Influence and Impact on Athlete Performance and Perception
Acronym: ANMATT
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University of Castilla-La Mancha (Other)
Responsible Party: Principal Investigator, Jose Luis Felipe, Senior Lecturer, University of Castilla-La Mancha
Allocation: Randomized | Model: Crossover | Masking: Single | Purpose: Basic Science
Other Study IDs: IGOID2
Record Dates: First submitted 2025-04-04; First posted 2025-04-22 (Actual); Last update posted 2025-04-22 (Actual); Status verified 2025-04

CONDITIONS: Artificial Turf; Athletic Performance and Injury Risk; Physical Fitness; Sports Equipment; Microplastics; Healthy
Keywords: Artificial Turf; Athletic Performance; Physical Fitness; Sports Equipment; Microplastics; Environmental Impact; Athlete Perception; Field Studies; Laboratory Testing; Synthetic Materials; Natural Materials; Polymer Infills; Durability; Safety; Functional Performance; Regulation Compliance; Third-Generation Turf; Football (Soccer)
MeSH Terms: interventions — CVD protocol

STUDY DESIGN:
Intervention Model Description: The study employs a crossover design to evaluate the impact of different artificial turf materials on athlete performance and perception. Participants, consisting of 30 amateur football players, will be randomly divided into groups. Each group will test six different types of artificial turf surfaces in a randomized order. The study includes a familiarization session followed by performance tests and perception assessments conducted over seven sessions. Each session lasts approximately two hours and includes various physical tests such as sprints, jumps, and small-sided games. The crossover design ensures that all participants experience each type of turf, allowing for comprehensive comparisons and minimizing bias. Data collected will be analyzed to determine the mechanical properties of the surfaces and their influence on athlete performance and perception.
Who Masked: Participant
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (6):
- Standard Turf (Experimental): articipants test the standard turf surface first, followed by the other surfaces in a randomized order.
  Interventions: Behavioral: Countermovement Jump (CMJ); Behavioral: Repeated Jump Test; Behavioral: Repeated Sprint Ability (RSA) Test; Behavioral: Maximum Sprint Test; Behavioral: Change of Direction (COD) Test; Behavioral: Shooting Test; Behavioral: Small side game test; Behavioral: Performance and Comfort Perception Questionnaire; Behavioral: Perceived Exertion Questionnaire
- Ecolastene Turf (Experimental): Participants test the Ecolastene turf surface, followed by the other surfaces in a randomized order.
  Interventions: Behavioral: Countermovement Jump (CMJ); Behavioral: Repeated Jump Test; Behavioral: Repeated Sprint Ability (RSA) Test; Behavioral: Maximum Sprint Test; Behavioral: Change of Direction (COD) Test; Behavioral: Shooting Test; Behavioral: Small side game test; Behavioral: Performance and Comfort Perception Questionnaire; Behavioral: Perceived Exertion Questionnaire
- Natural Turf (Experimental): Participants test the natural turf surface, followed by the other surfaces in a randomized order.
  Interventions: Behavioral: Countermovement Jump (CMJ); Behavioral: Repeated Jump Test; Behavioral: Repeated Sprint Ability (RSA) Test; Behavioral: Maximum Sprint Test; Behavioral: Change of Direction (COD) Test; Behavioral: Shooting Test; Behavioral: Small side game test; Behavioral: Performance and Comfort Perception Questionnaire; Behavioral: Perceived Exertion Questionnaire
- No Performance Infill Turf (Experimental): Participants test the turf surface without performance infill, followed by the other surfaces in a randomized order.
  Interventions: Behavioral: Countermovement Jump (CMJ); Behavioral: Repeated Jump Test; Behavioral: Repeated Sprint Ability (RSA) Test; Behavioral: Maximum Sprint Test; Behavioral: Change of Direction (COD) Test; Behavioral: Shooting Test; Behavioral: Small side game test; Behavioral: Performance and Comfort Perception Questionnaire; Behavioral: Perceived Exertion Questionnaire
- Natural Grass (Experimental): Participants test the hybrid turf surface, followed by the other surfaces in a randomized order.
  Interventions: Behavioral: Countermovement Jump (CMJ); Behavioral: Repeated Jump Test; Behavioral: Repeated Sprint Ability (RSA) Test; Behavioral: Maximum Sprint Test; Behavioral: Change of Direction (COD) Test; Behavioral: Shooting Test; Behavioral: Small side game test; Behavioral: Performance and Comfort Perception Questionnaire; Behavioral: Perceived Exertion Questionnaire
- Hybrid Turf (Experimental): Participants test the hybrid turf surface, followed by the other surfaces in a randomized order.
  Interventions: Behavioral: Countermovement Jump (CMJ); Behavioral: Repeated Jump Test; Behavioral: Repeated Sprint Ability (RSA) Test; Behavioral: Maximum Sprint Test; Behavioral: Change of Direction (COD) Test; Behavioral: Shooting Test; Behavioral: Small side game test; Behavioral: Performance and Comfort Perception Questionnaire; Behavioral: Perceived Exertion Questionnaire

INTERVENTIONS:
Behavioral: Countermovement Jump (CMJ) — Participants perform a vertical jump starting from a standing position, bending their knees to 90 degrees, and then jumping as high as possible. The height of the jump is measured using a laser measurement tool (OptoJump-Microgate, Optojump, Bolzano, Italy).
Behavioral: Repeated Jump Test — Participants perform repeated vertical jumps for 20 seconds, with the height of each jump measured using a laser measurement tool (OptoJump-Microgate, Optojump, Bolzano, Italy).
Behavioral: Repeated Sprint Ability (RSA) Test — articipants perform six 30-meter sprints with 20 seconds of rest between each sprint. Sprint times are measured using photocell timing gates (RaceTime, Microgate, Bolzano, Italy).
Behavioral: Maximum Sprint Test — Participants perform three maximum effort sprints over 40 meters. Sprint times and speeds are measured using 1080 motion analysis
Behavioral: Change of Direction (COD) Test — Participants perform a sprint with a change of direction, running 5 meters in one direction and then 5 meters at a 90-degree angle. The time to complete the test is measured.
Behavioral: Shooting Test — Participants perform a shooting test, aiming to hit a target with maximum speed. The speed of the shot is measured using radar.
Behavioral: Small side game test — Participants engage in a 5v5 small-sided game on a 600 m² field to simulate match conditions and assess performance in a game-like scenario.
Behavioral: Performance and Comfort Perception Questionnaire — Participants complete a questionnaire to assess their perception of performance and comfort on the surface, using a Visual Analogue Scale (VAS).
Behavioral: Perceived Exertion Questionnaire — Participants complete a questionnaire to assess their perceived exertion during the tests, using the Borg scale

SUMMARY:
This request pertains to a series of related projects on a common theme. Specifically, this set of projects aims to analyze the impact of new alternatives in materials and structures of artificial turf on athlete performance and perception, within the context of the elimination of microplastics as per Commission Regulation (EU) 2023/2055 of September 25, 2023. Third-generation sports artificial turf is notable for including performance infill (granules) that provide the necessary functionality and safety for sports practice. The vast majority of fields worldwide use materials that do not comply with the new European regulation, which has granted an eight-year moratorium. Therefore, there is little time to find new alternatives. The challenge lies not only in developing new structural solutions but also in understanding their impact on athletes. This issue is of high severity, as these sports facilities are the largest in terms of space and host the highest number of Physical Activity and Sports practitioners in Europe (mainly Football, Rugby, Hockey, and Padel).

For this reason, over the past year, the IGOID Group has requested various projects to cover all the necessary phases and nuances to address this issue.

The activities included in these projects are divided into two phases:

Phase 1: Evaluation of Sports Surfaces in the Laboratory (durability and surface-player and surface-ball interaction). Tests will be conducted on artificial turf samples constructed with SBR rubber (the main material to be replaced under the EU regulation), natural-origin infills, polymeric infills larger than 5 mm, and other infills. Initially, a market analysis and classification will be carried out, followed by laboratory tests. Across all projects, a minimum of 30 alternatives are expected to be analyzed.

Phase 2: Field Study. Tests will be conducted on a sample of athletes on constructed surfaces representing the different alternatives evaluated in Phase 1. Performance tests and a battery of assessments will be carried out to understand athlete perception. A sample of 30 athletes will be randomly divided into groups to perform different repetitions of the test batteries, covering a minimum of six different sports facilities.

ELIGIBILITY:
Inclusion Criteria: Gender: Male or female football players. Experience: Players who have played football for at least one full season prior to participating in the study.

Playing Level: Players who have played at the base or amateur level for at least 6 years.

Health Status: Players who do not have active or chronic injuries that could affect their ability to perform performance tests.

Willingness to Participate: Players who are willing to undergo performance tests and complete perception questionnaires.

Recent Injury History: Players who have not experienced significant injuries in the three months prior to the start of the study.

Medical Conditions: Players who do not have pre-existing medical conditions that could affect their ability to perform performance tests or endanger their health during the tests.

Medication: Players who are not taking medications that could affect their ability to perform performance tests.

Consent: Players who have signed an informed consent form to participate in the study and are willing to consistently follow the study protocols.

Age: Players between 20 and 30 years old (to obtain a more homogeneous sample). -

Exclusion Criteria: Recent Injury: Players who have experienced a significant injury in the last three months that required medical attention or could affect their ability to perform performance tests.

Chronic Illness: Players who have a chronic illness that could affect their ability to perform performance tests.

Medication: Players who are taking medications that could affect their ability to perform performance tests or could affect their understanding of the questionnaires and perception tools.

Medical History: Players who have a history of cardiovascular, pulmonary, or neurological disease.

Recent Surgery: Players who have had major surgery in the last six months that could affect their ability to perform performance tests.

Protocol Compliance: Players who are not willing or able to consistently follow the study protocols.

Disability: Players who have a physical or cognitive disability that could affect their ability to perform performance tests.

Consent: Players who have not signed an informed consent form to participate in the study.

Age: Players who do not meet the minimum and maximum age requirements to be included in the study.

-

Ages: 20 Years to 30 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 30 (Estimated)
Dates: Start 2025-09-01 (Estimated); Primary Completion 2025-12-30 (Estimated); Study Completion 2026-06-30 (Estimated)

PRIMARY OUTCOMES:
Performance Metrics on Different Surfaces | Sprint times: Measured at Baseline (Day 1) and Week 12. Jump heights: Measured at Baseline (Day 1) and Week 12. Agility: Measured at Baseline (Day 1) and Week 12.
  Sprint times (seconds): The time taken to complete a 20-meter sprint will be measured in seconds.
  Jump heights (meters): The height achieved during a vertical jump will be measured in meters.
  Agility (seconds): The time taken to complete an agility course will be measured in seconds.
Perception of Comfort and Performance | Immediately after each testing session on each surface
  Participants' subjective ratings of comfort and performance on each surface using a Visual Analogue Scale (VAS).Scale Details: The VAS will range from 0 to 100 mm, where:
  0 mm represents the lowest possible rating (e.g., "No comfort" or "Poor performance").
  100 mm represents the highest possible rating (e.g., "Maximum comfort" or "Excellent performance").
  Interpretation of Scores: Higher scores on the VAS indicate better outcomes, meaning higher comfort and better performance.

SECONDARY OUTCOMES:
Impact Absorption | Measured at Baseline (Day 1) during the initial evaluation of each surface.
  Measurement of impact absorption using the Artificial Athlete method (EN 14808: 2006). The results will be reported in kilonewtons (kN).
Rotational Resistance | Measured at Baseline (Day 1) during the initial evaluation of each surface.
  Measurement of rotational resistance using a traction device with a dynamometric key (EN 15301-1: 2008 and FIFA 2015) in N·m
Ball Rebound | Measured at Baseline (Day 1) during the initial evaluation of each surface.
  Measurement of ball rebound using a microphone (EN 12235: 2014 and FIFA 2015) in cm
Ball Roll | Measured at Baseline (Day 1) during the initial evaluation of each surface.
  Measurement of horizontal ball roll using a standardized angle ramp and photocells (FIFA 2015). In cm
Critical Fall Height | Measured at Baseline (Day 1) during the initial evaluation of each surface.
  Measurement of critical fall height using the Head Injury Criterion (HIC) (WR Regulation 22 2020) in cm
Perceived Exertion | Immediately after each testing session on each surface.
  Participants' ratings of perceived exertion during the tests using the Borg scale. The Borg scale ranges from 6 to 20, where:
  6 represents "No exertion at all". 20 represents "Maximal exertion". Interpretation of Scores: Higher scores on the Borg scale indicate higher levels of perceived exertion.
Vertical Deformation | Measured at Baseline (Day 1) during the initial evaluation of each surface.
  Measurement of vertical deformation using the Advanced Artificial Athlete method (FIFA 2015). The results will be reported in millimeters (mm).